CLINICAL TRIAL: NCT06710925
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of Monoclonal Antibody TNM001 Injection Against Respiratory Syncytial Virus in High-risk Infants
Brief Title: A Sudy to Evaluate the Efficacy and Safety of TNM001 in High-risk Infants
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhuhai Trinomab Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TNM001-302
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TNM001 (Experimental)
  Interventions: Biological: TNM001
- Placebo (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: TNM001 — single dose intramuscular injection
  Arms: TNM001
Biological: placebo — single dose intramuscular injection
  Arms: Placebo

SUMMARY:
This study is a Phase 3 randomized, double-blind, placebo-controlled study to evaluate the safety, efficacy, and immunogenicity of TNM001 in high-risk infants when entering their RSV season. Approximately 201 infants will be randomized in a ratio of 2:1 to receive TNM001 or placebo. All subjects will be followed for 270 days after dosing. This study will be conducted at approximately 20 sites in China.

ELIGIBILITY:
Inclusion Criteria:

* 1.High risk infants under 1 year of age who are entering their first RSV season at the time of screening.
* 2.Subject's legal representative(s) is(are) able to understand and comply with the requirements and procedures of the protocol,including scheduled visits and sample collection.
* 3.Subject is available to complete the follow-up period.

Exclusion Criteria:

* 1. Any fever (> 38.0°C) or acute illness within 7 days prior to randomization
* 2. History of RSV infection
* 3. Being hospitalized at the time of randomization
* 4. Currently receiving or expected to receive immunosuppressive therapy during the study period.
* 5. Renal impairment or hepatic dysfunction
* 6. Nervous system disease or neuromuscular disease
* 7. Known immunodeficiency including HIV, mother with HIV infection unless the child's infection has been excluded.
* 8. Known allergy history of immunoglobulin products, receipt or expected to receive immunoglobulins or blood products during the study period.
* 9.Receipt of RSV vaccine or mAb
* 10.Receiving blood products before randomization

Ages: 0 Weeks to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 201 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of medically attended LRTI due to RT-PCR confirmed RSV | 150 days post dose

CONTACTS AND LOCATIONS:
Overall Officials: Hanmin Liu, Principal Investigator — West China Second Hospital, Sichuan University; Enmei Liu, Principal Investigator — Children's Hospital of Chongqing Medical University
Locations (2):
- China (2):
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - Children's Hospital of Chongqing Medical University, Chongqing, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided